CLINICAL TRIAL: NCT03433196
Title: Randomized,Double Blind,Double Dummy, Multi-center Study of Efficacy and Safety of HS-25 Combination With Atorvastatin in Subjects With Hypercholesterolemia in Coronary Heart Diseases
Brief Title: Efficacy and Safety Study of the HS-25 Combination With Atorvastatin in Subjects With Hypercholesterolemia in Coronary Heart Diseases
Acronym: HS-25-III-02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang Hisun Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-25-III-02
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-02

CONDITIONS: Hypercholesterolemia in Coronaory Heart Disease
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind, Double dummy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-25 and Atorvastatin (Experimental): HS-25 20mg, Atorvastatin 10mg, Placebo of Atorvastatin 1 tablet
  Interventions: Drug: HS-25 and Atorvastatin
- Atorvastatin (Active Comparator): Atorvastatin 20mg, Placebo of HS-25 2 tablets
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: HS-25 and Atorvastatin — HS-25 20mg (2 tablets), Atorvastatin 10mg, Placebo of Atorvastatin 1 tablet oral, once daily
  Arms: HS-25 and Atorvastatin
Drug: Atorvastatin — Atorvastatin 20mg (2 tablets), Placebo of HS-25 2 tablets, oral, once daily
  Arms: Atorvastatin

SUMMARY:
To determine the efficacy of HS-25 (20mg) in reducing low density lipoprotein-cholesterol (LDL-C) levels after a 12-week period of treatment in combination with Atorvastatin in subjects with hypercholesterolemia and coronary heart diseases; To determine the safety of HS-25 (20mg) combination with Atorvastatin in subjects with hypercholesterolemia and coronary heart diseases

ELIGIBILITY:
Inclusion Criteria:

* Diet control for 14 weeks, Atorvastatin 10mg once daily for 6 weeks or above;
* The average of both qualifying values must be in the range of 2.07 mmol/L to 3.36 mmol/L. Run-in (Visit 2 and Visit 3) and the Visit 3 value must be within 12% of the value at Visit 2, higher or lower;
* Must meet the one of diseases as following:

  1. Subjects who have stable coronary heart disease;
  2. Subjects who diagnosed ischemic stroke in stable condition;
  3. Subjects who diagnosed as Diabetes mellitus

Exclusion Criteria:

* history of Severe Endiocrine disease (for example Thyroid function abnormal);
* History of advanced cancer
* Arrhythmias need to be treated by medications history of Hemorrhagic stroke;
* Cardiac dysfunction;
* Unstable ASCVD;
* History of organ transplant;
* Hypersensitive to HS-25 or place;
* uncontrolled or new diagnosed diabetes mellitus;
* HCV and HBsAg positive

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2016-06-07 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Percent change of LDL-C | 2,4,8,12 weeks
  Percent change from baseline in LDL-C after 2,4,8,12 weeks of double-blind treatment

SECONDARY OUTCOMES:
Percent change of Non-HDL-C | 2,4,8,12 weeks
  Percent change from baseline in Non-HDL-C after 2,4,8,12 weeks of double-blind treatment
Percent change of TC,TG,ApoB,ApoAI | 2,4,8,12 weeks
  Percent change from baseline in TC,TG,ApoB and ApoAI after 2,4,8,12 weeks of double-blind treat

CONTACTS AND LOCATIONS:
Overall Officials: Litong Qi, Principal Investigator — Peking University First Hospital